CLINICAL TRIAL: NCT04420520
Title: Prevalence of Molar Incisor Hypomineralization Among a Group of Egyptian Children in Fayoum Governorate Schools: A Cross Sectional Study
Brief Title: Prevalence of Molar Incisor Hypomineralization Among a Group of Egyptian Children in Fayoum Governorate Schools
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Snoussy Abo-alsaod, Pricipal Investigator, Cairo University
Other Study IDs: CEBD-CU-2020-05-13
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Molar Incisor Hypomineralization
Keywords: MIH
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determining the Prevalence of Molar Incisor Hypomineralization Among a Group of Egyptian Children in Fayoum Governorate Schools via clinical examination.

Participants from primary and preparatory schools in Fayoum governorate will be included in the study and Clinical examination will be carried out in the school laboratory or an empty class, in day light for both genders.

Teeth will be cleaned gently using gauze and wet with saliva during examination. A disposable diagnostic set (mirror, probe) will be used for each patient where mirrors will be used for proper visualization especially for maxillary teeth. Blunt explorers will be used to aid in tactile sensation if needed, as during the differentiation between rough and smooth enamel edges and/or during the inspection of the caries extent if it exists. No diagnostic radiographs will be taken.

The results of the study will be regularly monitored by the supervisors who will have full access to these results.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance for participation in the study.
* Eruption of four first permanent molars.
* Eruption of four permanent maxillary and mandibular incisors.
* Both genders.

Exclusion Criteria:

* Uncooperative children.
* Children with orthodontic appliances.
* Children with systemic diseases which may affect teeth development.
* Children suffering from any other type of enamel defect as enamel hypoplasia and amelogenesis imperfecta.

Ages: 6 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: Egyptian children in Fayoum governorate schools.
Sampling Method: Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2020-09-20 (Estimated); Primary Completion 2021-04-20 (Estimated); Study Completion 2021-05-20 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Molar Incisor Hypomineralization | Through study completion, an average of 1 year
  Prevalence of Molar Incisor Hypomineralization done via clinical examination using a disposable diagnostic set in the school laboratory or an empty class, in day light.